CLINICAL TRIAL: NCT02295709
Title: Cervical Transforaminal Injection of Steroids Guided by Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Dongping Du, Pain Management Center, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-46
Record Dates: First submitted 2014-11-16; First posted 2014-11-20 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Cervical Radiculopathy
Keywords: ultrasound; cervical Transformational Epidural Steroid Injection
MeSH Terms: conditions — Radiculopathy | interventions — Dexamethasone; Injections; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- USNR steroid injection (Experimental): the patient who are treated with steroid (dexamethasone) injection through selected cervical spinal nerve block approach guided by ultrasound and C arm.
  Interventions: Procedure: SNR steroid (dexamethasone) injection; Drug: Dexamethasone; Device: Ultrasound; Radiation: C arm
- UCTF steroid injection (Experimental): the patients who are treated with steroid (dexamethasone) injection through cervical transforaminal approach guided by ultrasound and C arm.
  Interventions: Procedure: CTF steroid (dexamethasone) injection; Drug: Dexamethasone; Device: Ultrasound; Radiation: C arm
- XCTF steroid injection (Experimental): the patients who are treated with steroid (dexamethasone) injection through cervical transforaminal approach guided only by C arm.
  Interventions: Procedure: CTF steroid (dexamethasone) injection; Drug: Dexamethasone; Radiation: C arm

INTERVENTIONS:
Procedure: SNR steroid (dexamethasone) injection — deliver steroids (dexamethasone) into spinal nerve root with the guidance of ultrasound.
  Device: Ultrasound (S-Nerve; SonoSite, Bothell, Wash), Probe 9L (6 MHz, SonoSite, Bothell, Wash)
  Arms: USNR steroid injection
Procedure: CTF steroid (dexamethasone) injection — deliver steroids (dexamethasone) into spinal epidural space with the guidance of ultrasound.
  Device: Ultrasound (S-Nerve; SonoSite, Bothell, Wash), Probe 9L (6 MHz, SonoSite, Bothell, Wash)
  Arms: UCTF steroid injection; XCTF steroid injection
Drug: Dexamethasone — One of the most efficient steroids
  Other Names: DXM
Device: Ultrasound — Ultrasound (S-Nerve; SonoSite, Bothell, Wash), Probe 9L (6 MHz, SonoSite, Bothell, Wash)
  Arms: UCTF steroid injection; USNR steroid injection
Radiation: C arm — the needle position will be re-confirmed by C arm C arm (Philips Healthcare, Best, the Netherlands）

SUMMARY:
Cervical transforaminal epidural steroid injections (TFESI) are indicated in cervical radicular pain resistant to conservation therapy, by which steroids can be delivered into anterior epidural space surrounding target spinal nerve roots to help alleviate pain in the upper limb or neck. Cervical TFESI is traditionally commended to perform with guidance of fluoroscopy or CT. As fluoroscopy can not monitor the injection route whether it pass vessel or not, many serious neurological complications caused by inadvertent intra-arterial injection have been reported2. Here, the investigators will introduce a novel cervical TFESI guided by ultrasound, which incidence of inadvertent vessel injury or injection might be lower than those guided by fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* evidence of a cervical radiculopathy involving 1 spinal nerve of at least 1 month's duration refractory to medical treatment
* symptoms of cervical pain radiating to the upper limb
* and signs of altered sensations, ab- normal reflexes, or motor weakness caused by degenerative spondylosis and/or disk herniation as documented at CT or MR imaging and a current mean pain VAS score of six.

Exclusion criteria:

* evidence of vertebral fracture, tumor, or infection of the cervical spine
* treatment with cervical corticosteroid injections within the past 3 months
* coagulopathy
* allergy to iodinated contrast media.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
change of pain severity rated on a Visual Analog Scale (VAS) | 1 day before, 1day after, 1week after and 4 weeks after the intervention

SECONDARY OUTCOMES:
change of neck actives rated on Neck Disability Index (NDI) | 1 day before, 1day after, 1week after and 4 weeks after the intervention
change of medication use rated on Medication Quantitative Scale (MQS) | 1 day before, 1day after, 1week after and 4 weeks after the intervention